CLINICAL TRIAL: NCT07014254
Title: Therapeutic Study of 177Lu-CTR-FAPI-targeted Nuclear Drugs in Advanced Metastatic Digestive Malignancies
Brief Title: Therapeutic Study of 177Lu-CTR-FAPI in Advanced Metastatic Digestive Malignancies
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: KY20252131-C-1
Record Dates: First submitted 2025-05-22; First posted 2025-06-10 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-05

CONDITIONS: Pancreatic Ductal Adenocarcinoma (PDAC); Adenocarcinoma of the Stomach; Colorectal Cancer Metastatic; Neuroendocrine Tumor (NET)
Keywords: 177Lu-CTR-FAPI
MeSH Terms: conditions — Neuroendocrine Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 177Lu-CTR-FAPI nuclide-targeted therapy (Experimental): 177Lu-CTR-FAPI nuclide-targeted therapy in patients with advanced tumours lacking effective treatments
  Interventions: Drug: 177Lu-CTR-FAPI nuclide-targeted therapy

INTERVENTIONS:
Drug: 177Lu-CTR-FAPI nuclide-targeted therapy — Fasting, special diets, or other specific preparations are not required on the day of 177Lu-CTR-FAPI administration. Patients were given 4 mg ondansetron 30 minutes before treatment to prevent nausea and vomiting. The radiopharmaceutical 177Lu-CTR-FAPI (200 ± 10% mCi) was diluted with 100 mL of 0.9% saline and given slowly by intravenous infusion over 20-30 minutes (flow rate 200 ml/h). Symptoms and vital signs were monitored before and after treatment. The treatment regimen was planned for a maximum of 3 courses of treatment, with 4-8 weeks between each cycle

SUMMARY:
This was a single-centre, single-arm, non-blinded, prospective study using 20 patients with advanced metastatic GI malignancies recruited to treat patients with advanced metastatic GI malignancies with 177Lu-CTR-FAPI to assess the safety of 177Lu-CTR-FAPI in advanced metastatic GI malignancies; this included radiation therapy dosimetry and initial treatment Determination of Effectiveness

ELIGIBILITY:
Inclusion Criteria:

* 1. voluntary participation in this study and signing of informed consent;
* 2. age 18-75 years (both 18 and 75 years);
* 3. ECOG (Eastern Cooperative Oncology Group) physical status score: 0-1;
* 4.Advanced metastatic gastrointestinal malignancies with high FAP expression: e.g. neuroendocrine tumours (NET G2, G3), neuroendocrine carcinomas (NEC), pancreatic ductal adenocarcinomas (PDAC), gastric adenocarcinomas, colorectal carcinomas, intrahepatic cholangiocarcinomas (ICC), and squamous carcinomas of the oesophagus. All of the above should be confirmed by 68Ga-FAPI PET/CT with high FAP expression (criterion: more than 50% of lesions with SUVmax ≥10). 5.
* 5. Disease status: locally advanced unresectable or metastatic lesions confirmed by imaging (CT/MRI/PET-CT); at least 1 measurable lesion (RECIST 1.1 criteria).
* 6. good major organ function, i.e. the following criteria are met (no blood components, cell growth factors are allowed within 14 days prior to the first dose)

  1. Creatinine clearance ≥ 50 ml/min (calculated according to the Cockcroft-Gault formula) or serum creatinine ≤ 150 μmol/L;
  2. Urine protein <2+; if urine protein ≥2+, then 24-hour urine protein quantification must show <2 g of protein;
  3. White blood cell count ≥ 2 × 109/L;
  4. Absolute neutrophil count (ANC) ≥ 1.5 × 109/L;
  5. Platelets ≥ 75 × 109/L;
  6. Haemoglobin ≥ 8.0 g/dL;
  7. Serum albumin ≥ 30 g/L.
  8. Total bilirubin ≤ 3 × ULN;
* 7. Women of childbearing age who undergo a blood pregnancy test within 72 h prior to treatment need to be excluded from pregnancy and must be non-lactating and willing to use a highly effective method of contraception for the duration of the trial and for 6 months after completion of treatment. For men, agreement to use a highly effective method of contraception or to have been surgically sterilised during the study and for 4 months after the end of treatment.

Exclusion Criteria:

* 1. Disease-related:

  1. Combination of other malignancies (except non-melanoma skin cancer or radical tumours without recurrence within 5 years);
  2. Presence of central nervous system metastases or carcinomatous meningitis;
  3. Uncontrolled cancer pain (requiring long-term high-dose opioids) or cachexia (≥20% weight loss in 6 months);
  4. Diabetes mellitus (fasting blood glucose > 2 x ULN) that is not well controlled with optimal medical supportive therapy;
  5. Accompanied by poorly controlled plasmapheresis, including pleural fluid, ascites, and pericardial effusion; controlled with treatment and stable (asymptomatic, not requiring interventional therapy, and stable on imaging) for ≥2 weeks may be included;
  6. Severe urinary incontinence, hydronephrosis, severe voiding dysfunction or the need for an indwelling urinary catheter for any reason;
  7. Subjects with uncontrolled cardiac clinical symptoms or disease, including but not limited to: i) NYHA class 2 or higher heart failure; ii) unstable angina; iii) myocardial infarction within 1 year prior to enrolment; iv) left ventricular ejection fraction (LVEF) <50%; v) clinically significant supraventricular or ventricular arrhythmias requiring treatment or intervention;
  8. Co-occurring active hepatitis B (HBV-DNA testing is required for HBsAg-positive individuals with HBV DNA ≥500 IU/mL or 2500 copies/mL), and hepatitis C (HCV-Ab-positive and above the lower limit of detection of the analytical method);
  9. Persons known to have acquired immunodeficiency syndrome (AIDS) or human immunodeficiency virus (HIV) testing positive. Persons with active syphilis infection.
* 2. Treatment related

  1. Radiotherapy within 4 weeks or previous radiotherapy to >25% of the bone marrow area;
  2. Received systemic anti-tumour therapy such as chemotherapy, immunotherapy, targeted therapy within 4 weeks;
  3. Treatment with surgery (biopsy puncture, non-anti-tumour surgical operations such as ERCP may be excluded), radiofrequency ablation or cryoablation, interferon, transcatheter arterial embolisation (TAE) or transcatheter arterial chemoembolisation (TACE) within 12 weeks;
  4. Prior FAP-targeted therapy (e.g., FAPI-PRRT, anti-FAP antibody drugs);
  5. Presence of contraindications to radionuclide therapy (e.g., myelodysplastic syndrome, extensive bone metastases with bone marrow failure).

     Comorbidities and Risks:
  6. Previous antineoplastic therapy resulting in toxicity that has not recovered to grade ≤1 according to the NCI-CTCAE v5.0 classification (with the exception of lowered lymphocyte counts, alopecia, and the indicators mentioned in the inclusion criteria, and with the exception of partially tolerable chronic grade 2 toxicity, in the judgement of the investigator).
* 3. Other exclusions

  1. History of allergy to peptide radiopharmaceuticals;
  2. Inability to co-operate with long-term follow-up (e.g., mental illness, geographical constraints, etc.);
  3. Refusal of contraception by pregnant or lactating women or patients of childbearing age.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-06-20 (Estimated); Primary Completion 2028-04-30 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
ORR | End of treatment (12 weeks)
  Objective mitigation rate
DCR | End of treatment (12 weeks)
  Disease control rate

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Nuclear Medicine,Xijing Hospital, Fourth Military Medical University, Xi'an, China, Xi'an, Shaanxi Province Recruiting, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No